CLINICAL TRIAL: NCT05197179
Title: A Randomized, Double-Blind, Placebo-Controlled, Bridging Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of FB2001 in Healthy Subjects
Brief Title: A Bridging Study of FB2001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB2001-101
Record Dates: First submitted 2021-12-16; First posted 2022-01-19 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — FB2001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Single-dose A (Other): A single dose A of FB2001 or placebo will be administered by intravenous (IV) infusion
  Interventions: Drug: FB2001; Other: FB2001 placebo
- Single-dose B (Other): A single dose B of FB2001 or placebo will be administered by intravenous (IV) infusion
  Interventions: Drug: FB2001; Other: FB2001 placebo
- Multiple-dose A (Other): Dose A of FB2001 or placebo will be administered by intravenous (IV) infusion once daily for 5 consecutive days
  Interventions: Drug: FB2001; Other: FB2001 placebo
- Multiple-dose B (Other): Dose B of FB2001 or placebo will be administered by intravenous (IV) infusion twice daily for 5.5 consecutive days
  Interventions: Drug: FB2001; Other: FB2001 placebo
- Single-dose C (Other): A single dose C of FB2001 or placebo will be administered by intravenous (IV) infusion
  Interventions: Drug: FB2001; Other: FB2001 placebo

INTERVENTIONS:
Drug: FB2001 — Subjects will be administered with FB2001 by intravenous (IV) infusion
  Other Names: DC402234
Other: FB2001 placebo — Subjects will be administered with FB2001 by intravenous (IV) infusion

SUMMARY:
In the first human clinical trial conducted in the United States, single and multiple dosing of FB2001 in multiple dose groups were partially completed，and FB2001 demonstrated good safety and tolerability. The bridge study of FB2001 will be conducted in China to evaluated the safety and PK of FB2001 in healthy Chinese population. This is a randomized, double-blind, placebo-controlled study of single and multiple dosing.

DETAILED DESCRIPTION:
Coronaviruses belong to the genus of coronavirus of the family coronaviruses. The viruses of the coronavirus genus are positive-sense single-stranded RNA viruses with envelopes, which are approximately 80-160 nm in diameter. Their genetic material is the largest among all RNA viruses and can infect both humans and animals. Coronaviruses can cause respiratory, intestinal, hepatic, and nervous system diseases of different severities. A total of 7 coronaviruses have been found, in which HCoV-229E, HCoV-OC43, HCoV-NL63 and HCoV-HKU1 mainly lead to mild and self-limiting upper respiratory tract infections in infected humans, such as common cold; two new types of β-coronaviruses have emerged in the past 12 years, namely severe acute respiratory syndrome (SARS-CoV) and Middle East respiratory syndrome (MERS-CoV), and these two viruses can cause severe human diseases.

In the first human clinical trial conducted in the United States, single and multiple dosing of FB2001 in multiple dose groups were partially completed，and FB2001 demonstrated good safety and tolerability. The bridge study of FB2001 will be conducted in China to evaluated the safety and PK of FB2001 in healthy Chinese population. This study is a randomized, double-blinded, placebo-controlled, ascending dose to evaluate the pharmacokinetics, safety and tolerability of FB2001 for injection afer a single and multiple dose administrations in healthy subjects. A total of 40 healthy subjects are planned to be enrolled. Each group will include 8 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults who are between 18 and 60 years old inclusive
2. Weigh at least 45kg, with a BMI of 19 to 30 kg/m2 inclusive
3. No serious underlying disease
4. Subjects should have normal (or abnormal but not clinically significant) laboratory results per the PI's judgement, including complete blood count, biochemistry, coagulation indices and urinalysis
5. Subjects should have a normal (or abnormal but not clinically significant) ECG and chest X-ray at screening
6. Current non-smokers and those who have not smoked within the last 6 months. This includes the use of cigarettes, e-cigarettes, and nicotine replacement products.
7. Female subjects should have negative results in serum pregnancy test at screening and negative urine pregnancy test at screening.
8. Agree to have no parenting plan during the study period and for 3 months after administration, and be able to use highly effective contraceptive measures, such as:

   * Complete abstinence (e.g. as the preferred lifestyle)
   * Intrauterine device (IUD)
   * Female barrier method: cervical or uterine cap with spermicidal agent
   * Tubal sterilization
   * Vasectomy for male subjects or partners
   * Hormone-containing contraceptives
   * Levonorgestrel implant
   * Progesterone injection
   * Oral contrceptives (combined or progesterone alone)
   * Vaginal contraceptive ring
   * Transdermal contraceptive patch
9. Willing to cooperate and be able to participate in the study, comply with all requirements of the program, and sign informed consent. .

Exclusion Criteria:

1. HIV antibody positive;
2. HBsAg positive;
3. HCV antibody positive;
4. Syphilis spirochetes antibody positive;
5. History of tuberculosis or lung disease as reported by subject;
6. Subject has severe cardiovascular disease, neurological disease, hematological disease, infectious disease, mental disorder, liver disease, gastrointestinal disease, endocrine disease, immune disease or kidney disease, or has a history of the above diseases, or other symptoms known to interfere with the absorption, distribution, metabolism, or excretion of the medicine, or other conditions that the investigator believes will increase the risk of the subject and might interfere with the study conduct and results interpretations;
7. Female subjects who are pregnant, lactating or have pregnancy plans and cannot contracept as required;
8. Subjects who participated in any other clinical study within 3 months prior to screening;
9. Subjects with known allergic reactions to the study drug or its excipients;
10. Subjects donated or lost ≥ 400 mL 3 months prior to the administration of study drugs; or subjects donated (including aphersis donation) or lost ≥ 200 mL 1 month prior to the administration;
11. Subjects who have taken any drug that inhibits or induces hepatic drug-metabolizing enzymes (e.g., inducers: barbiturate, carbamazepine, phenytoin, glucocorticoid, omeprazole; inhibitors: antidepressants like selective serotonin reuptake inhibitor (SSRI), cimetidine, diltiazem macrolides, nitroimidazoles, sedative-hypnotic drugs, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration; or subjects who have taken any prescription, over-the-counter, and herbal medications other than those listed above within 14 days prior to administration;
12. Alcoholics or regular drinkers within 3 months, i.e., those who comsume more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of liquor with 40% ABV or 150 mL of wine), or those who have a positive result in breath alcohol test;
13. Use of any medication, including prescription, over-the-counter, vitatmins, herbal and/or mineral supplements, dietary supplements (and/or grape fruit juice) within 14 days prior to the first administration, in the Investigator's judgment, which may influence study results or subjects' safety;
14. Any other clinical condition that, in the inverstigator's judgement, would potentially compromise study compliance or the abilityti evaluate safety and efficacy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of FB2001 after a single and multiple dose administrations in healthy subjects | Day1 - Day 29
  The safety and overall tolerability assessments will be evaluated based on:
  * Incidence of Treatment-Emergent Adverse Events (TEAEs) and Adverse reactions (ADR)
  * Incidence of grade 3 and 4 AEs/ADRs
  * Incidence of SAE
  * Incidence of drug-related serious adverse events
Pharmacokinetic parameter (AUC0-τ) | Day1 - Day 6
  Pharmacokinetic outcome measures: Estimate of steady state AUC0-τ for single and multiple dose administration of FB2001
Pharmacokinetic parameter (Cmax) | Day1 - Day 6
  Pharmacokinetic outcome measures: Estimate of steady state Cmax for single and multiple dose administration of FB2001

CONTACTS AND LOCATIONS:
Overall Officials: Yun Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China